CLINICAL TRIAL: NCT03085251
Title: Clinical System Accuracy Evaluation With OneTouch® Verio Flex Blood Glucose Monitoring System (BGMS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDT-1653-LI
Record Dates: First submitted 2017-03-15; First posted 2017-03-21 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Self-Testing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood glucose measurement (Experimental)
  Interventions: Device: Blood glucose monitoring systems for self-testing (BGMS)

INTERVENTIONS:
Device: Blood glucose monitoring systems for self-testing (BGMS) — Measurement procedure
  * Subjects will be asked to wash and dry their hands before the measurements.
  * The measurement procedure for each reagent system lot of a BGMS will be as follows:
  * Study personnel will collect a capillary blood sample from the subject's fingertip by skin puncture.
  * Duplicate measurements on the sample will be consecutively performed with 2 test meters using reagent system units from the same vial / package.
  * Capillary blood for measurements with all 3 test strip lots and for both comparison measurements will be taken from the same finger puncture.
  * The sample will be applied to the reagent system units following specifications in the manufacturer's labelling.
  Other Names: OneTouch® Verio Flex

SUMMARY:
The objective of this study is the evaluation of system accuracy based on EN ISO 15197:2015 (ISO 15197:2013), clause 6.3 in which accuracy requirements and applicable test procedures for blood glucose monitoring systems intended for self-monitoring of blood glucose by patients are stipulated. ISO 15197:20132 was harmonized with the regulations of the European Union as EN ISO 15197:2015. This harmonization had no impact on the requirements and procedu¬res in ISO 15197:2013; changes were made to the foreword and an informative annex. In this study, system accuracy evaluation will be performed for OneTouch® Verio Flex (LifeScan Europe) on behalf of LifeScan Scotland Limited (customer) with three different reagent system lots.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, with type 1 diabetes, type 2 diabetes (or subjects without diabetes)
* Signed informed consent form
* Minimum age of 18 years
* Subjects are legally competent and capable to understand character, meaning and consequences of the study.
* If blood glucose values < 80 mg/dl or > 300 mg/dl shall be measured after short term alteration in insulin therapy:
* Male or female with type 1 diabetes and intensified insulin therapy or insulin pump therapy.
* Signature of subjects to document consent with these procedures on informed consent form.

Exclusion Criteria:

* Pregnancy or lactation period
* Severe acute disease (at the study physician's discretion)
* Severe chronic disease with potential risk during the test procedures (at the study physician's discretion)
* Current constitution that compromises the subject's capability to participate in the study (at the study physician's discretion)
* Being unable to give informed consent
* < 18 years
* Legally incompetent
* Being committed to an institution (e.g. psychiatric clinic)
* Language barriers potentially compromising an adequate compliance with study procedures
* Dependent on investigator or sponsor
* If blood glucose values < 80 mg/dl shall be measured after short term alteration in insulin therapy (concentration category 2), subjects with type 1 diabetes, suffering from:
* Coronary heart disease
* Condition after myocardial infarction
* Condition after cerebral events
* Peripheral arterial occlusive disease
* Hypoglycemia unawareness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2017-04-03 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
System accuracy criteria | For each subject, the experimental phase has an expected duration of up to 6 hours
  Based on EN ISO 15197:2015 (ISO 15197:2013) (E), the BGMS shall meet both of the following criteria:
  Criterion A: 95 % of the measured glucose values shall fall within either ± 15 mg/dl (0.83 mmol/l) of the average comparison measurement result at glucose concentrations < 100 mg/dl (5.55 mmol/l) or within ± 15 % at glucose concentrations ≥ 100 mg/dl (5.55 mmol/l).
  Each lot shall pass acceptability criterion A. Criterion B: 99 % of individual glucose measured values shall fall within zones A and B of the Consensus Error Grid (CEG) for type 1 diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Baden-Wurttemberg, Germany